CLINICAL TRIAL: NCT01428466
Title: Dermal Safety Study of GSK2585823 (Clindamycin 1%-Benzoyl Peroxide 3% Gel) With Healthy Japanese Male and Female Subjects
Brief Title: Japanese Phase 1 Study of GSK2585823
Acronym: JPN P1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 114849
Record Dates: First submitted 2011-06-16; First posted 2011-09-05 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- GSK2585823 (Experimental): external preparation
  Interventions: Drug: GSK2585823
- Benzoic peroxide 3% (Active Comparator): external preparation
  Interventions: Drug: Benzoyl peroxide 3%
- Benzoic peroxide 5% (Active Comparator): external preparation
  Interventions: Drug: Benzoyl peroxide 5%
- Vehicle (Placebo Comparator): external preparation
  Interventions: Other: Vehicle

INTERVENTIONS:
Drug: GSK2585823 — CLDM1%/BPO3%
  Arms: GSK2585823
Drug: Benzoyl peroxide 3% — Benzoyl peroxide 3%
  Arms: Benzoic peroxide 3%
Drug: Benzoyl peroxide 5% — Benzoyl peroxide 5%
  Arms: Benzoic peroxide 5%
Other: Vehicle — placebo
  Arms: Vehicle

SUMMARY:
This is a randomized, single-center, partial-blind study to evaluate the dermal irritation potential and to detect photo-toxicity and photo-allergy potential of GSK2585823, Benzoyl peroxide BPO 5% gel, Benzoyl peroxide 3% gel, vehicle gel and negative control (distilled water) applied using Finn-Chambers® by single and 7-day repeat patch test in 20 Japanese healthy male and female volunteers. Finn-Chambers containing no investigational product will be applied in the same manner.

Safety will also be assessed by measurement of vital signs, electrocardiograms, safety laboratory data and review of adverse events.

DETAILED DESCRIPTION:
Each subjects will be applied the adequate amount of GSK2585823, Benzoyl peroxide 3%, Benzoyl peroxide 5%, placebo (Vehicle) and negative control (distilled water) using Finn Chambers on Scanpor (the tape for the patch test which Finn Chamber® put on the Scanpor® tape in advance) on their upper back at same time for the simple patch test and the photo patch test. The empty Finn Chamber® will also be applied at the same time. The position of application for each product (including empty Finn Chamber®) will be randomized The position of application for each subjects will be same for the simple patch test and the photo patch test.

For the simple patch test, dermal condition will be assessed up to 48 hours after removal of the Finn-Chambers®. After removing the Finn-Chambers®, the skin areas will be gently wiped with wet absorbent cotton before the first evaluation at 30 minutes.

For the photo patch test, two sets of Finn-Chambers® will be applied to the skin. Twenty-four hours after the single application or the last application of the repeat dosing, a set of Finn-Chambers® will be removed. The skin areas will be gently wiped and exposed to 6.0 J/cm2 of ultraviolet A. The other set of Finn-Chambers® are covered to avoid ultraviolet A exposure to serve as un-irradiated control when photo-allergy is assessed 30 minutes after ultraviolet A exposure. After the assessment, the skin areas will be covered with empty Finn-Chambers® for additional 24 hours to prevent further exposure to light. Photo-toxicity will be assessed 24 and 48 hours after the ultraviolet A exposure.

Assessment of Simple Patch test

1. The dermatologist will examine the planned application sites and skin reactions at the application sites, and make assessments at the following time points according to the criteria proposed by the patch test study group in Japan.

   <Single application phase> Day 1: just before application Day 3: 30 minutes after removal of study medication (48.5 hours after application) Day 4: 24 hours after removal of study medication (72 hours after application) <Repeat application phase> Day 5: just before application Days 6-11: every 24 hours (30 minutes after removal; about 23.5 hours after application). This result will be used only for safety assessment and not for calculation of irritation index.

   Day 12: 30 minutes after removal of last study medication (24.5 hours after the last application) Day 13: 24 hours after removal of last study medication (48 hours after the last application) Day 14: 48 hours after removal of last study medication (72 hours after the last application)

   Assessment Criteria Proposed by Patch Test Study Group in Japan No visible reaction(-); 0 Minimal visible erythema(±); 0.5 Erythema(+); 1 Erythema + edema(++); 2 Erythema + edema + papules + vesicles(+++); 3 Erythema bullosum (++++); 4
2. The dermatologist will examine that application site on Day 4 for single application phase and Day 14 for repeat application phase to determine whether the symptom is an allergic reaction or not.

Assessment of Photo Patch Test

1. The scorer (dermatologist) will examine the planned application sites and skin reactions at the application sites, and make assessments at the following time points according to the criteria proposed by the patch test study group of Japan Dermatology Society].

   <Single application phase> Day 1: just before application Day 3: 24 hours after irradiation (48 hours after application) Day 4: 48 hours after irradiation (72 hours after application) <Repeat application phase> Day 5: just before application Day 13: 24 hours after removal of last study medication (48 hours after the last application) Day 14: 48 hours after removal of last study medication (72 hours after the last application)
2. The dermatologist will examine the irradiation sites 30 minutes after irradiation (about 24.5 hours after the start of application) on Day 2 (single) and to determine whether there is photo-urticaria or not.
3. 30 minutes after irradiation to determine whether there is photo-urticaria or not. Then, 24 and 48 hours after irradiation, the skin reactions at the irradiation sites will be compared with the corresponding non-irradiation site for photo patch test, using the criteria showing in Table 1 and the photo-toxicity of each investigational product will be assessed according to the following criteria.

Assessment Criteria for Photo-toxicity No reaction or similar to the non irradiation site; - Slightly stronger than the non irradiation site; ± Definitely stronger than the non irradiation site; + 2 ranks stronger than the non irradiation site according to the criteria in Japan; ++ 3 ranks stronger than the non irradiation site according to the criteria in Japan; +++

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as determined by a responsible and experienced physician.
2. Japanese healthy male and female subjects aged between 20 and 45 years of age inclusive, at the time of signing the informed consent.
3. Asparate aminotransferase(AST), Alanine aminotransferase(ALT) and total bilirubin < Upper level of normal range
4. Non-smoker (never smoked or not smoking for >6 months with <10 pack years history (Pack years = (cigarettes per day smoked/20) x number of years smoked)).
5. Body Mass Index (BMI) within the range =>18.5 to < 25.0 kg/m2 at screening
6. A female subject is eligible to participate if she is of:

   * Non-childbearing potential.
   * Child-bearing potential and agrees to use one of the contraception methods from screening to the follow up examination.
7. Capable of giving written informed consent.
8. Single QTcB < 450 msec at screening

Exclusion Criteria:

1. A positive test for syphilis, Hepatitis B surface antigen or positive Hepatitis C antibody, HIV antibody and HTLV-1 result at screening.
2. A positive for urine drug screening.
3. History of regular alcohol consumption within 6 months of the study defined as:

   -an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 350 mL of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
4. The subject has participated in a clinical study with an investigational or a non-investigational drug or device during the previous 4 months.
5. The subject planned to concurrently participate in another clinical study or post-marketing study.
6. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days prior to the first application of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
7. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
8. The subject has donated a unit of blood ">400 mL" within the previous 4 months or ">200 mL" within the previous 1 month.
9. Pregnant females as determined by positive urine hCG test at screening or prior to dosing.
10. Lactating females.
11. Unwillingness or inability to follow the procedures outlined in the protocol.
12. Subject is mentally or legally incapacitated.
13. Subjects with clinically significant skin diseases which may contraindicate participation, or interfere with test site evaluations, including psoriasis, eczema, atopic dermatitis, acne, dysplastic nevi, or other skin pathologies.
14. Subjects with a history of hypersensitivity or idiosyncratic reaction to benzoyl peroxide, clindamycin, lincomycin or any study medication components or requiring significant concomitant medications or with diseases affecting evaluation of study medication
15. Subjects with scars, moles, other blemishes or tattoos, darkened skin or excessive hair on the utilised area of the mid or upper back which would interfere with grading the test sites
16. Within six months (oral) or 2 weeks (topical) prior to and during the study, subjects must not be treated with retinoids.
17. For one month (systemic) or 2 weeks (topical) before and during the study, subjects not to be treated with corticosteroids or any other medication that could interfere with study results.
18. Subjects with sunburn or suntan on test area of mid or upper back
19. Subjects with considerable exposure to sunlight, including sunlamps, on test area of mid or upper back
20. Subjects with inherent sensitivity to sun or history of photosensitivity

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-11-18 (Actual); Primary Completion 2011-02-15 (Actual); Study Completion 2011-02-15 (Actual)

PRIMARY OUTCOMES:
Dermal irritancy (simple patch test) | Participants will be followed for the duration of hospital stay, an expected average of 22 days.
Photo allergy and toxicity (Photo patch test) | Participants will be followed for the duration of hospital stay, an expected average of 22 days.

SECONDARY OUTCOMES:
Photo-toxicity and photo-allergy potential (photo-patch test) | Participants will be followed for the duration of hospital stay, an expected average of 22 days.
Safety and tolerability endpoints: adverse events, blood pressure, heart rate, 12-lead ECG, clinical laboratory safety tests | Participants will be followed for the duration of hospital stay, an expected average of 22 days.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Nakahara N, Nohda S, Hirama T. Dermal safety of GSK2585823 in healty Japanese subjects. [J Clin Therapeut Med]. 2012;(September):867-876.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 114849 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114849?search=study&study_ids=114849#rs
- Available data/document: Individual Participant Data Set: 114849 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114849 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114849 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114849 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register